CLINICAL TRIAL: NCT02082600
Title: Effects of Sleep Deprivation on Blood Hormones and Inflammatory Status After Exercise Induced-muscle Damage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Hanna Karen Moreira Antunes, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2010070050
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Sleep; Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep deprivation (Experimental): Exercise induced-muscle damage protocol followed by 60h of sleep deprivation (two nights) and one night of normal sleep (rebound).
  Interventions: Other: Sleep deprivation
- Normal sleep (Experimental): Exercise induced-muscle damage protocol followed by 3 nights of normal sleep
  Interventions: Other: Normal sleep

INTERVENTIONS:
Other: Sleep deprivation — This group will perform 24 sets of 10 maximum repetitions of eccentric contractions for quadriceps and than will keep awake for 60 hours (2 nights), followed by 1 night of sleep, all inside the lab. During whole protocol, it will be collected several blood samples for evaluation of hormones, cytokines and muscle damage parameters. It will be also evaluated isometric strength and pain.
  Other Names: Sleep and muscle recovery
  Arms: Sleep deprivation
Other: Normal sleep — This group will perform 24 sets of 10 maximum repetitions of eccentric contractions for quadriceps and and will be able to sleep the 3 nights. During whole protocol, it will be collected several blood samples for evaluation of hormones, cytokines and muscle damage parameters. It will be also evaluated isometric strength and pain.
  Arms: Normal sleep

SUMMARY:
The aims of this study are examine the effects of sleep deprivation in muscle recovery after a maximum eccentric resistance exercise session performed on an isokinetic dynamometer (24 series of 10 repetitions). The sample will consist of 10 men, sedentary, clinically healthy, aged between 20 and 31 years old. Two experimental groups will be developed: EXE-SLEEP, in which subjects will perform the exercise protocol (~18:00-19:00) and will be subject to normal period of sleep for 3 nights; EXE-TOTAL, in which subjects will perform the same exercise protocol and will be sleep deprived for 60 hours, followed by one night of sleep rebound.

DETAILED DESCRIPTION:
The blood parameters analyzed will be:

* Creatine kinase and myoglobin: before, immediately after, 2, 4, 12, 24, 36, 48, and 60 hours after exercise protocol.
* Total and free testosterone, IGF-1, and cortisol: before, immediately after, 2, 4, 12, 24, 36, 48, and 60 hours after exercise protocol. Moreover, from 19:00 of the second day to 19:00 of the third day it will be collected blood samples every 2 hours.
* GH: during the second night, GH will be evaluated every 1 hour, from 23:00 to 07:00.
* TNF-alfa, IL-6, IL-1 beta, IL-10, and IL-1ra: before, immediately after, and 2 hour after exercise, as well every 4 hours from 19:00 of the second day to 19:00 of the third day.

It will be evaluated isometric strength every 12 hours, as well visual analog scale of pain.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* sedentary
* sleep duration between 6-8 hours peer night

Exclusion Criteria:

* smokers
* use vitamin supplements, like C and E
* drink two doses of alcohol/day or > 4 doses in one occasion
* use of anti-inflammatory drugs
* antilipidemic drugs
* anemia
* muscle or joint diseases
* cardiovascular diseases
* diabetes
* renal diseases
* sleep disturbances
* breathing disorders

Ages: 20 Years to 31 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in isometric strength | Before exercise, immediatly after, 12, 24, 36, 48, and 60 hours after exercise induced-muscle damage

SECONDARY OUTCOMES:
Area Under Curve for serum total and free testosterone, IGF-1, and cortisol | Blood samples will be collected every 2 hours, for 24 hours.

OTHER OUTCOMES:
Area Under Curve for serum pro and anti-inflammatory cytokines | Blood samples will be collected every 4 hours, for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tulio Mello, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Associação Fundo de Incentivo à Pesquisa, São Paulo, São Paulo, Brazil